CLINICAL TRIAL: NCT05743335
Title: A PHASE 1 STUDY to ASSESS the SAFETY and IMMUNOGENICITY of a BROADLY PROTECTIVE MRNA VACCINE JCXH-221 AGAINST SARS-CoV-2 INFECTION and DISEASES
Brief Title: A Phase 1 Study to Assess the Safety and Immunogenicity of JCXH-221, an MRNA-based Broadly Protective COVID-19 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immorna Biotherapeutics, Inc. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JCXH-221-001
Record Dates: First submitted 2023-02-22; First posted 2023-02-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Infectious Disease
Keywords: mRNA Vaccine; COVID vaccination; Healthy subjects
MeSH Terms: conditions — COVID-19; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: 2 age groups will be enrolled in parallel for Phase 1 (18-64 age group and 65+ age group).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational product (Experimental): Patients randomized to this arm will be given the investigational product (JCXH-221).
  Interventions: Biological: JCXH-221
- Placebo (Placebo Comparator): Patients randomized to this arm will be given a placebo vaccine.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: JCXH-221 — Participants will be randomized to either placebo or JCXH-221 for Phase 1. For Phase 2, participants will either be randomized to JCXH-221 or a FDA approved Active comparator.
  Arms: Investigational product
Other: Placebo — Participants will be randomized in Phase 1 to either JCXH-221 or placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about, test, and compare JCXH-221 in healthy volunteers. The main aims to answer are:

* To assess the safety and tolerability of the JCXH-221 vaccine in healthy adult subjects
* To identify an optimal dose for the JCXH-221 vaccine in healthy adult subjects
* To assess the humoral immunogenicity of the JCXH-221 vaccine in healthy adult subjects
* To characterize the cellular immunogenicity of the JCXH-221 vaccine in healthy adult subjects

Participants for Phase I will be randomized to either JCXH-221 or placebo.

DETAILED DESCRIPTION:
This is a phase 1 study looking to enroll a total of 72 patients.

For phase 1, two cohorts will be explored (18-64 age group and 65+ age group) for a total of 72 subjects. The subjects will be enrolled and randomized to either placebo or JCXH-221. A low dose of JCXH-221 will be explored vs placebo for each age group first.

ELIGIBILITY:
Main Inclusion Criteria

* Sex: Male or female; female subjects may be of childbearing potential, of nonchildbearing potential, or postmenopausal.
* Age: 18 years of age or older, at screening.
* Status: Healthy subjects.
* Subjects must have completed the full doses for primary vaccination with an approved SARS-CoV-2 vaccine and may have received booster dose(s), with the last vaccination (can be 2nd dose of primary vaccination or booster dose) having occurred at least 4 months prior to enrollment.

Main Exclusion Criteria

* Current or prior symptomatic or asymptomatic SARS-CoV-2 infection confirmed by an approved or authorized rapid antigen test on Day 1 or within 4 months prior to Day 1.
* Subjects with significant exposure (as defined by current CDC guidance) to someone with laboratory confirmed SARS-CoV-2 infection or COVID-19 with the past 14 days prior to the Screening visit.
* Subjects with fever or signs of acute infection at the time of enrollment and vaccination.
* Subjects who are taking medications that may prevent or treat COVID-19.
* Subjects who received convalescent serum or prior therapeutic antibodies against SARS-CoV-2 within 4 months before Day 1.
* Subjects with history of myocarditis or pericarditis, or with AEs after mRNA vaccination that are in nature and severity beyond the common AEs expected and necessitating medical intervention.
* Subjects with active or suspected immunosuppression, immunodeficiency, or autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
SAE frequency | Day 1- Day 365 (12 months)
  Frequency of serious adverse events (SAEs) characterized by type, severity, duration, and drug relationship, from Day 1 (dosing day) until follow-up completion
Injection site reaction | Day 1- Day 8 (7 days)
  Solicited local reactions at the injection site characterized by frequency, severity, and duration, recorded up to 7 days after dosing (Day 8)
Solicited systemic reaction frequency | Day 1- Day 8 (7 days)
  Solicited systemic reactions characterized by frequency, severity, duration, and drug relationship, recorded up to 7 days after dosing (Day 8)
AE frequency | Day 1- Day 29 (28 days)
  Adverse events (AEs), including unsolicited AEs, characterized by frequency, severity, duration, and drug relationship, for up to 28 days after dosing (Day 29)
Unsolicited treatment-emergent AE frequency | Day 1- Day 29 (28 days)
  The proportion of subjects with at least 1 unsolicited treatment-emergent AE occurring up to 28 days after dosing (Day 29)
Medical AE frequency | Day 1- Day 365 (12 months)
  Medically attended AEs (MAAEs) characterized by frequency, severity, duration, and drug relationship, from Day 1 until follow-up completion

SECONDARY OUTCOMES:
SARS-CoV-2 antibody levels | Day 1- Day 181 (~6 months)
  Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)-specific serum neutralizing antibody levels against ancestral and variant SARS-CoV-2 strains as compared to baseline (Day 1 predose) at 7, 14, and 28 days after dosing, and 2, 4, and 6 months after dosing:
  * Geometric mean titers (GMTs) at each time point
  * Geometric mean-fold rise (GMFR) from before vaccination to each subsequent time point after vaccination
  * Seroresponse rate (SRR) defined as the proportion of subjects achieving ≥4-fold rise from before vaccination to each subsequent time point after vaccination
SARS-CoV-2 anti-receptor antibody levels | Day 1- Day 181 (~6 months)
  SARS-CoV-2 anti-receptor binding domain (RBD) antibody levels as compared to baseline (Day 1 predose) at 7, 14, and 28 days after dosing, and 2, 4, and 6 months after dosing
  * Geometric mean concentrations (GMCs) at each time point
  * GMFR from before vaccination to each subsequent time point after vaccination
  * SRR defined as the proportion of subjects achieving ≥4-fold rise from before vaccination to each subsequent time point after vaccination

OTHER OUTCOMES:
T-cell responses | Day 1- Day 181 (~6 months)
  T-cell responses to vaccine-encoded antigen and antigen-specific memory B cells and plasmablasts in peripheral blood mononuclear cells determined by enzyme-linked immunosorbent spot (ELISpot) assays, as compared to baseline (Day 1 predose) at 14 days and 6 months after dosing (Day 15 and Month 6)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Velocity Clinical Research, Hallandale, Florida
  - Velocity Clinical Research, Savannah, Georgia
  - Velocity Clinical Research, Lincoln, Nebraska
  - Velocity Clinical Research, Cedar Park, Texas

IPD SHARING:
Plan to Share IPD: No